CLINICAL TRIAL: NCT03069079
Title: Investigation of Dental Health in Children With Neutrophil Defects: A Clinical Study
Acronym: GOSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COCR0004; 011374 (Registry Identifier: QMUL R and D); 15/LO/1090 (Other: UK REC)
Record Dates: First submitted 2017-01-17; First posted 2017-03-03 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2016-12

CONDITIONS: Primary Immune Deficiency Disorder; Periodontitis
Keywords: primary immunodeficiency; dental health; neutrophil defect; periodontitis
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non surgical Periodontal therapy (Experimental): All children will be offered an oral hygiene and tooth scaling and polishing session. For children affected by periodontal disease, subgingival debridement will also be performed according to needs, with the aim to disrupt the subgingival biofilm responsible for the onset and progression of the periodontal pathology. This can be accompanied, when appropriate, by the use of local anaesthesia and adjunctive antimicrobials (systemic or locally applied subgingivally), according to the clinical presentation and the child's medical conditions. In addition, when required, nitrous oxide sedation (NOS) could be used before treatment.
  Caries will be treated as necessary (shared care with the general dental practitioners / community dental services). Children with mucosal lesions requiring treatment will be given a letter for their GDP suggesting referral to a collaborating expert in Oral Medicine (Prof. Stephen Porter).
  Interventions: Procedure: Oral hygiene advice, non surgical periodontal treatment

INTERVENTIONS:
Procedure: Oral hygiene advice, non surgical periodontal treatment — For children affected by periodontal disease, oral hygiene advice, non surgical periodontal treatment will also be performed according to needs. This can be accompanied, when appropriate, by the use of local anaesthesia and adjunctive antimicrobials (systemic or locally applied subgingivally), according to the clinical presentation and the child's medical conditions. Accurate supra- and sub-gingival removal of calculus and dental plaque will be performed both with ultrasonic and/or manual instruments. The necessary sub-gingival debridement will be performed in 1 to 4 visits (either full mouth treatment, half-mouth treatment or quadrant-wise treatment) depending on patient preference and practical considerations, using manual (Gracey curettes, Hu-Friedy) and ultrasonic devices (EMS). .

SUMMARY:
Title: Investigation of neutrophil defects associated with periodontal disease and tooth loss in children. A clinical study.

Objectives: The primary objective of this study is:

* To investigate presence of periodontal disease and response to periodontal treatment in children affected by neutrophil defects

The secondary objectives of this study are:

* To investigate presence of other dental diseases in children affected by neutrophil defects
* To assess oral microbiological and inflammatory parameters in children affected by neutrophil defects

Primary outcomes: The primary outcomes are (a) presence of periodontal disease as assessed by clinical factors: probing pocket depth, attachment level, bleeding on probing and radiographic bone loss) (b) microbiological and host response factors: detected in periodontal pockets and gingival crevicular fluid and (c) response to treatment

Study sample: Children affected by neutrophil defects and meeting outlined inclusion and exclusion criteria

Number of participants: 50 children

Study design: This is a longitudinal treatment study. All participants will attend for 4-7 visits during the study as outlined below:

* Screening visit (visit 1): consent procedure, dental examination, saliva and plaque sampling
* Baseline visit (visit 2):, detailed periodontal examination, dental radiographs, sampling of gingival crevicular fluid and, if appropriate scaling, polishing and oral hygiene instructions
* Non-surgical periodontal treatment (visit 3A to 3D, max 4 sessions): oral hygiene instructions and supra- and sub-gingival debridement (under local anaesthesia if necessary)
* Follow-up Visit (visit 4, 4th to 7th visit) (six months following treatment): detailed dental examination, oral hygiene instructions, sampling of saliva, subgingival plaque and gingival crevicular fluid, tooth scaling and polishing.

DETAILED DESCRIPTION:
1. BACKGROUND Primary immunodeficiency diseases (PIDs) are a group of rare inherited disorders that are estimated to affect approximately 1 in 2,000 children. In PIDs there is an intrinsic defect in the human immune system, such as a failure to produce enough antibodies to fight infection, or a failure in the cellular defences against infection . These conditions usually manifest themselves early in life and are often life-threatening. Rarer, severe forms of PIDs present in childhood with serious infections and are often associated with additional autoimmune and inflammatory complications. Periodontal diseases are inflammatory diseases of the gingivae (gums) due to an imbalance in the host response to subgingival bacteria and are associated with destruction of the supporting tissues of the teeth and early loss of the dentition and masticatory function. While periodontitis and its non-destructive partner condition, gingivitis (reversible plaque-induced gingival inflammation), are very common, the prevalence of periodontitis in the primary dentition and in the second decade of life appears very low, ranging from 0.1% to 1%. This prevalence increases dramatically in children affected by PIDs, to the point that periodontitis is considered a common feature of syndromic genetic conditions due to single gene defects affecting the host response, such as leukocyte adhesion deficiency (LAD), severe congenital neutropenia, cyclic neutropenia and Chediak-Higashi syndrome. Children with defects in neutrophil activity seem particularly susceptible to develop severe periodontitis, due to the important defensive role of neutrophils against periodontopathogenic bacteria. In such cases, both primary and permanent dentitions are affected, with a devastating effect on mastication, aesthetics and quality of life, also owing to the lack of reliable restorative solutions. Furthermore, oral diseases (in particular periodontitis) may also provide an additional systemic inflammatory burden for these subjects. This could occur since periodontal bacteria have been shown to enter the systemic circulation from inflamed gum tissues even during normal tooth brushing, have been found in atheromatous plaques and in the amniotic fluid of pregnant women.

   The treatment of periodontitis involves a non-specific reduction of the bacterial load below the gingival margin, achieved by oral hygiene instructions and non-surgical periodontal therapy (NSPT). More advanced cases need antibiotics, surgical treatment or extractions. In children with PID the response to this treatment is highly variable and the presence of periodontitis often leads to early tooth loss, adding to the poor quality of life of sufferers. Incorporation of periodontal screening has been advocated for early diagnosis and treatment of periodontal diseases in all children and especially for children with neutrophil defects, in order to prevent disease progression and tooth loss. However, most published papers on periodontitis in children with immunodeficiencies are case reports or familial observations or reviews. Therefore, there's a lack of well-designed studies investigating both the prevalence of periodontitis and oral diseases in general in children with neutrophil defects and their response to treatment. In particular, it is not clear which factors determine the onset of periodontitis in a subset of children with PID. Such factors may range from the composition of the subgingival microbiota, the immunological reaction against these bacteria, to the inflammatory response in the periodontium. A better understanding of the causative factors may help in early diagnosis and treatment, reducing the burden on affected children.
2. AIMS AND OBJECTIVES

   The hypotheses behind this study are that:

   i) Specific microbiological and host response parameters dictate severity of periodontal diseases and associated risk of early tooth loss in children suffering from neutrophil defects ii) Periodontal treatment in children with neutrophil defects and periodontitis can lead to an improvement in their oral health (reduction in periodontal pockets and bleeding scores), which would reduce their risk of tooth loss and potentially improve their future quality of life.

   Therefore, the aims of this study are to offer specialist periodontal assessment and treatment to children with neutrophil defects, to determine the impact of neutrophil defects upon gingival health and to assess their response to periodontal therapy. This will facilitate the development of novel therapeutic management pathways specific for these conditions, and will determine whether there is a need for specific care protocols with a consequent improvement in tooth retention, quality of life and systemic health.
   * The primary objective of this study is:

     - To investigate presence of periodontal disease and response to periodontal treatment in children affected by neutrophil defects
   * The secondary objectives of this study are:

     * To investigate presence of other dental diseases in children affected by neutrophil defects
     * To assess oral microbiological and host response parameters in children affected by neutrophil defects.
3. STUDY DESIGN 3.1 Overall study plan This is an exploratory longitudinal study. Fifty children affected by neutrophil defects potentially affecting the periodontium will be identified from subjects attending the Immunology and Haematology clinics at Great Ormond Street Hospital (GOSH), following a medical examination. All children will undergo a dental examination by a qualified dentist currently completing specialist training in periodontology. Children will also provide samples of gingival crevicular fluid (GCF) and subgingival plaque. Following the baseline, non-surgical periodontal therapy will be provided as necessary and participants will be followed-up and re-examined up to 6 months after treatment.
4. STUDY POPULATION 4.1 Participant Selection Fifty children affected by neutrophil defects and under care at Great Ormond Street Hospital (GOSH) and meeting the inclusion criteria will participate in the study. Most children attend GOSH regularly (at least 6-monthly) for review/treatment planning appointments (seen by Dr Ancliff or Dr Worth). The parents/guardians of potentially suitable children will be initially contacted by letter prior to their attendance at GOSH. Every invitation will be followed up by a telephone call to discuss any issues and enquiry about willingness to participate. When possible, upon parents' agreement about study participation, patients could be enrolled and undergo the screening visit on the same day as their routine GOSH visit (this would save on extra travel for patients living outside London). Alternatively, they will be offered another appointment. All the study visits will take place at GOSH. QMULwill only serves as the sponsor and coordinating centre for this study. .
5. STUDY VISITS Study visits include baseline, non-surgical periodontal therapy and follow-ups. All visits will be carried out at Great Ormond Street Hospital.

   5.1 Visit 1 (Screening) o Informed consent

   o Collection of data on clinical and laboratory diagnosis, time of diagnosis, previous and current systemic treatment and on any previous dental treatment

   o Basic Periodontal Examination (BPE) and assessment of caries (DMFT) and mucosal diseases

   o Saliva and plaque sample
   * Clinical photographs
   * Treatment plan All children found to have BPE scores of 1 (gingival bleeding), 2 (presence of calculus), 3 or 4 (presence of gingival pockets) will be offered the possibility to enter the treatment phase of the study (from visit 2 onwards), which will be provided at GOSH. Children found not to be affected by periodontal diseases will be offered the possibility to be seen at GOSH for visit 2 only, if they wish so.

   5.2 Visit 2 (Baseline and first treatment session- ± 28 days) o Recording of any adverse events (AE or concomitant medication)
   * Full periodontal examination including collection of periodontal measurements (and dental radiographs if appropriate)
   * Gingival crevicular fluid (GCF) sample
   * Session of tooth scaling, oral hygiene and polishing

   All children found to require further treatment will need to attend an additional 1 to 4 treatment sessions at GOSH as detailed below:

   5.3 Visit 3A to 3D (treatment, within 2 months of visit 1, from 1 to 4 visits) Update medical history, check adverse events, non-surgical periodontal therapy (maximum 4 sessions): oral hygiene instructions and supra- and sub-gingival debridement.

   5.4 Visit 4 (last follow-up, 6 months after last treatment visit ± 21 days) Update medical history, check adverse events, dental examination and collection of periodontal measurements, perform oral hygiene instructions, sampling of saliva, subgingival plaque and gingival crevicular fluid, tooth scaling and polishing (if needed).

   5.5 Medical and dental history A complete medical and dental history will be obtained during screening and confirmed during the baseline visit. Information on previous medical tests and status of current treatment will be obtained by the treating GOSH physician. The histories will include demographic background information, ethnicity, systemic and dental status information.

   5.6 Concomitant medications All concomitant medications will be recorded throughout the study.

   5.7 Periodontal examination At the screening visit, a Basic Periodontal Examination (BPE) will be performed, consisting of gentle probing between teeth and gums on index teeth (UR6, UR1, UL6, LL6, LL1 and LR6 or URd,URc,ULd,LLD,LLc,LRd) to identify presence of gum disease. A number between 0 (health) and 4 (gingival pocket>5mm) will be recorded for each quadrant. The dmft/ DMFT (decayed missing filled teeth) index will be used for recording caries experience. Mucosal status will be investigated by recording presence of ulcers, blisters, white patches, speckled areas and masses. Saliva samples and plaque samples will be collected. At the baseline visit, a calibrated dental examiner will perform a more detailed assessment, consisting of collection of full-mouth measurements of probing pocket depth (PPD), clinical attachment level (CAL), gingival bleeding on probing gingival crevicular fluid sampling and assessment of plaque levels (simplified visible biofilm index).

   5.8 Dental sampling A series of samples will be collected from the patients' oral cavity (sample of saliva, GCF and subgingival plaque biofilm). GCF will be taken by gentle insertion of 4 paper-strips in the gingival crevice of the mesio-buccal aspect of 4 teeth (3 first molars and 1 incisor). Subgingival plaque will be collected by the examiners following gentle insertion of a curette at the base of 3 first molars and 1 first incisor sites (one in each quadrant). In case of absence of permanent molars, the samples will be collected from the second deciduous molars. The 4 subgingival samples will be pooled together.

   5.9 Definition of periodontal disease

   Following the periodontal examination, children will be diagnosed as:

   - Healthy: no attachment loss (measured as no CAL>3mm or CAL>3mm in <2 non-adjacent teeth) and no/minimal gingival inflammation (measured as <15 sites bleeding on probing)

   - Gingivitis: no attachment loss (measured as no CAL>3mm or CAL>3mm in <2 non-adjacent teeth) and presence of gingival inflammation (≥15 sites bleeding on probing)

   - Periodontitis: attachment loss (measured as CAL>3mm in ≥2 non-adjacent teeth)

   5.10 Dental radiographs If a BPE code 3 or more is detected, bite-wings or long cone parallel periapical radiographs (more indicated for a BPE of 4) using Rinn holders will be taken to detect marginal bone levels, according to clinical needs. The distance between coronal and apical bone levels and cemento-enamel junction will be analysed as described previously, also taking into account age of the patient, tooth eruption stage and presence of primary, mixed or permanent dentition. Radiographs will then be digitized for future analysis using an image-analysis software.

   5.11 Non-surgical periodontal treatment All children will be offered an oral hygiene and tooth scaling and polishing session. For children affected by periodontal disease, subgingival debridement will also be performed according to needs, with the aim to disrupt the subgingival biofilm responsible for the onset and progression of the periodontal pathology. This can be accompanied, when appropriate, by the use of local anaesthesia and adjunctive antimicrobials (systemic or locally applied subgingivally), according to the clinical presentation and the child's medical conditions. In addition, when required, nitrous oxide sedation (NOS) could be used before treatment. NOS is a safe and widely-used technique in paediatric dentistry. It is administered by inhalation via a nasal mask and is used to reduce dental anxiety along with behaviour management techniques. There are very few contra-indications. It is not suitable for patients who have nasal congestion or severe dental anxiety. NOS will be conducted following the guidelines by Standards for Conscious Sedation in the Provision of Dental Care and appropriate clinical consent forms will be obtained before its use.

   Accurate supra- and sub-gingival removal of calculus and dental plaque will be performed both with ultrasonic and/or manual instruments. The necessary sub-gingival debridement will be performed in 1 to 4 visits (either full mouth treatment, half-mouth treatment or quadrant-wise treatment) depending on patient preference and practical considerations, using manual (Gracey curettes, Hu-Friedy) and ultrasonic devices (EMS). Caries will be treated as necessary (shared care with the general dental practitioners / community dental services). Children with mucosal lesions requiring treatment will be given a letter for their GDP suggesting referral to a collaborating expert in Oral Medicine (Prof. Stephen Porter).
6. Missing data The inclusion of very young subjects in the present study introduces the risk of missing data, owing to the difficulty in data and sample collection in some children (due to their unwillingness to be examined or sampled). The Investigators will endeavor to complete data and sample collection with minimal discomfort to each subject. However, should dental and periodontal examination not be achievable, the subjects will be exited from the study. Once the main variable outcome of the study (presence of periodontal disease by means of collection of BPE) is recorded, the subject will not be excluded from analysis, even if some of the other data are not collected. For example, if a child tolerated periodontal probing (hence collection of BPE) but refuses to provide a plaque sample, he/she will still be included in the study until the last visit. The final study analyses and report/publications will take into account possible missing data and reasons why they were not collected.

5.7 Repeatability Prior to initiation of the study, the designated examiner will participate in a training and repeatability exercise. For the repeatability exercise, the examiner will score 5 subjects for PPD and REC and then perform repeated examinations of the same subjects on the same day after at least 15 minutes separation. Upon completion of all measurements, intra-examiner repeatability for PPD measurements will be assessed. The reproducibility of the examiner will be tested using the Bland-Altman approach and by calculating Lin's concordance correlation coefficient. A co-efficient of repeatability less than ± 2 mm in 95% of the cases is considered acceptable.

5.8 Laboratory analyses Samples will initially be stored at -70° to -80° for analysis. Microbiological analysis will involve next generation sequencing of the 16S rRNA metagenome at QMUL. GCF samples will be eluted and will undergo analysis of inflammatory markers as described before.

9. PARTICIPANTS' COMPLETION AND WITHDRAWAL 9.1Reasons for withdrawal

Participants will be informed that they have the right to withdraw from the study at any time for any reason, without prejudice to their medical care. The investigator also has the right to withdraw participants from the study for any of the following reasons:

* Occurrence of an unacceptable adverse event/illness
* Participant/parent/guardian request
* Protocol violations
* Administrative reasons
* Failure to return for follow-up
* General or specific changes in the Participant's condition unacceptable for further treatment in the judgment of the investigator

9.2 Completion/Withdrawal Procedures At the time of withdrawal, all study procedures outlined for the end of study visit should be concluded. The primary reason for a participant's withdrawal from the study is to be recorded on the CRF.

10. ADVERSE EVENT REPORTING 7.1 Adverse Events (AEs) An adverse event includes any noxious, pathological or unintended change in anatomical, physiological or metabolic functions as indicated by physical signs, symptoms and/or laboratory changes occurring in any phase of the clinical study, whether associated with the study or not. This includes exacerbation of pre-existing conditions or events, inter-current illnesses, drug interaction or the significant worsening of the disease under study. For all adverse events, the investigator must pursue and obtain information adequate both to determine the outcome of the adverse event and to assess whether it meets the criteria for classification as a serious adverse event requiring immediate notification to the sponsor or its designated representative. For all adverse events, sufficient information should be obtained by the investigator to determine the causality of the adverse event.

Clinically significant symptoms following NSPT include those that are outside a normally accepted range (as judged by the clinician). This would include:

* Excessive or progressively increasing pain or discomfort
* Excessive swelling
* Signs of infection (e.g. suppuration)
* Excessive bleeding

Moreover we shall record if the participants take any drugs as a result of these adverse events.

7.2 Serious Adverse Events definition

A serious adverse event or serious adverse drug reaction is any untoward medical occurrence at any dose which:

* results in death
* is life-threatening (immediate risk of death)
* requires participant hospitalization or prolongation of existing hospitalization
* results in persistent or significant disability/incapacity
* results in congenital anomaly/birth defect.

Medical and scientific judgment should be exercised in determining whether an event is an important medical event. An important medical event may not be immediately life-threatening and/or result in death or hospitalization. However, if it is determined that the event may jeopardize the participant and may require intervention to prevent one of the other outcomes listed in the definition above, the important medical event should be reported as serious.

7.3 Reporting of Serious Adverse Events Because of the need to report to health authorities all suspected unexpected serious adverse reactions (SUSARs) in a timely manner, it is vitally important that the investigator reports immediately any adverse events which would be considered serious. Any serious adverse event (including death) due to any cause, which occurs during the course of this clinical study, whether or not related to the study, must be reported immediately to the Principal Investigator or its designee.

7.4 Reporting period The nature of each individual adverse event, date and time of onset, duration, severity and relationship to treatment and corrective treatment must be established by the investigator and recorded in the CRF. Adverse events will be recorded following signing of the first consent form up to the last study visit. Any serious adverse event occurring any time after the reporting period must be promptly reported if a causal relationship to the investigational product is suspected and all SUSARs will be followed up until resolution.

8 STATISTICAL PROCEDURES 6.1 Sample size estimation A convenience sample of 50 children (based on current estimation of numbers of children with neutrophil defects seen yearly at GOSH) is proposed for this study, since no formal power calculation could be performed owing to the lack of similar studies in the literature. However, hypothesising that subgingival presence of bacterium A.actinomycetemcomitans at baseline could discriminate between responders and non-responders to periodontal treatment (difference 0.5mm ± 0.5 mm mean clinical attachment gain), 41 children (including 20% drop-outs) who undergo periodontal therapy would give 80% power to prove or disprove this hypothesis.

6.2 Statistical analysis All data derived from the study will be anonymised and entered in a dedicated database. The initial plan of analysis will describe the prevalence of periodontal diseases in the study cohort (divided by medical diagnosis). Appropriate summary statistics will be determined separately for affected and non-affected subjects. Differences in demographic and systemic parameters (diagnosis, current treatment) between affected and non-affected subjects will be assessed by the two-sample t-test or Mann-Whitney test as appropriate. Explorative logistic regression analyses will be performed to detect the effect of microbiological and inflammatory parameters (e.g. presence of periodontopathogenic bacterium A.actinomycetemcomitans or cytokine concentrations in the GCF) on groups, taking into account that many children may be on long-term antimicrobial therapy. Response to therapy will be assessed by comparing clinical periodontal parameters at baseline and follow-ups by random effects analysis taking time points as repeated measures. This will be then associated to patients' demographics, compliance and microbiological and inflammatory factors.

7 ADMINISTRATIVE REQUIREMENTS 9.1 Good clinical practice The study will be conducted in accordance with the International Conference on Harmonisation (ICH) for Good Clinical Practice (GCP) and the appropriate regulatory requirement(s). Essential clinical documents will be maintained to demonstrate the validity of the study and the integrity of the data collected. Master files should be established at the beginning of the study, maintained for the duration of the study, and retained according to the appropriate regulations.

9.2 Ethical considerations The study will be conducted in accordance with ethical principles founded in the Declaration of Helsinki. The Research Ethics Committee will review all appropriate study documentation in order to safeguard the rights, safety, and well-being of the participants. The study will be conducted only at sites where Research Ethics Committee approval has been obtained. The protocol, informed consent, advertisements (if applicable), written information given to the participants, safety updates, progress reports, and any revisions to these documents will be provided to the Research Ethics Committee by the investigator.

9.3 Participant Information and Informed Consent During the first screening session and the enrolment visit, written informed consent will be obtained from all participants/guardians/parents. The method of obtaining and documenting the informed consent and the contents of the consent will comply with ICH-GCP and all applicable regulatory requirement(s).

9.4 Participant confidentiality In order to maintain participant privacy, all CRFs, study reports and communications will identify the participant by initials and the assigned participant number. The participant's confidentiality will be maintained and will not be made publicly available to the extent permitted by the applicable laws and regulations.

9.5 Protocol compliance The investigator will conduct the study in compliance with the protocol and given approval/favorable opinion by the Research Ethics Committee and the appropriate regulatory authority(ies). Changes to the protocol will require written Research Ethics Committee approval/favourable opinion prior to implementation, except when the modification is needed to eliminate an immediate hazard(s) to participants.

9.6 Study monitoring Monitoring and auditing procedures developed by the investigator will be followed, in order to comply with GCP guidelines. On-site checking of the CRFs for completeness and clarity, cross-checking with source documents, and clarification of administrative matters will be performed. The study will be monitored by a clinical trial coordinator or its designee.

9.7 Case report form completion Case report forms will be completed for each study participant. It is the investigator's responsibility to ensure the accuracy, completeness, and timeliness of the data reported in the participant's CRF. Source documentation supporting the CRF data should indicate the participant's participation in the study and should document the dates and details of study procedures, adverse events and participant status.

The investigator, or designated representative, should complete the CRF pages as soon as possible after information is collected, preferably on the same day that a study participant is seen for an examination, treatment, or any other study procedure. Any outstanding entries must be completed immediately after the final examination. An explanation should be given for all missing data. The investigator must sign and date the Investigator's Statement at the end of the CRF to endorse the recorded data.

9.8 Premature closure of the study This study may be prematurely terminated, if in the opinion of the investigator there is sufficient reasonable cause. Written notification, documenting the reason for study termination, will be provided to the investigator by the terminating party.

Circumstances which may warrant termination include, but are not limited to:

* Determination of unexpected, significant, or unacceptable risk to participants
* Failure to enter participants at an acceptable rate
* Insufficient adherence to protocol requirements
* Insufficient data

9.9 Complaints and indemnity

* Complaints. In the event of complaint about the conduct of the study, the hosting NHS- Great Ormond Street Hospital for Children NHS Foundation - complaints policy should apply as the research subject is recruited through an NHS Trust.
* Indemnity QMUL holds insurance against claims from participants for harm caused by their participation in this clinical study. Participants may be able to claim compensation if they can prove that QMUL has been negligent. However, if this clinical study is being carried out in a hospital, the hospital continues to have a duty of care to the participant of the clinical study. QMUL does not accept liability for any breach in the hospital's duty of care, or any negligence on the part of hospital employees. This applies whether the hospital is an NHS Trust or otherwise.

ELIGIBILITY:
Inclusion Criteria

Each participant must meet the following inclusion criteria to be enrolled in the study:

1. Age 4-16 years
2. Diagnosis of one of the following neutrophil defects (as confirmed by the treating physician):

   * Disorders of neutrophil numbers

     * Cyclic neutropenia
     * Congenital neutropenia
     * Severe Congenital Neutropoenia
     * X-linked Neutropoenia
   * Disorders of neutrophil function

     * Leucocyte Adhesion Defect s
     * Other neutrophil disorders/ undefined neutrophil disorders (functional defects demonstrated on testing but genetic basis not yet known)
   * Combined immunodeficiency syndromes

     * Wiskott Aldrich Syndrome
     * Hyper IgM Syndrome
     * Chediak Higashi Syndrome
     * Undefined combined immunodeficiency (functional defects demonstrated on testing but genetic basis not yet known)
3. Participants/parents/guardians willing to sign the informed consent Exclusion Criteria Participants will not be eligible for participation in the study if unwilling to be examined or unable to return for follow-up appointments.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2016-12; Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth | At baseline only (0 months)
  Measurement periodontal pocket depth at baseline (in millimetres, mm)
Attachment level | At baseline only (0 months)
  Measurement of attachment level at baseline (in millimetres, mm)
Bleeding on probing | At baseline only (0 months)
  Proportion of bleeding sites on probing at baseline (in percentage, %)
Radiographic bone loss | At baseline only (0 months)
  Proportion of bone loss in relation to total root length at baseline. (in percentage, %)
Microbiological assay | At baseline only (0 months)
  Microbiological analysis with next generation sequencing of the 16s rRNA metagenome at baseline. (Proportion of specified microbes present in sample at baseline)
GCF | At baseline only (0 months)
  Gingival crevicular fluid inflammatory markers (Proportion specified inflammatory markers present in sample at baseline)

SECONDARY OUTCOMES:
Response to treatment: Probing pocket depth | From baseline (0 months) to follow-up (24 months)
  Change in periodontal pocket depth at baseline to follow-up (in millimetres, mm)
Response to treatment: Attachment level | From baseline (0 months) to follow-up (24 months)
  Change in proportion of bleeding sites on probing at baseline to follow-up (in percentage, %)
Response to treatment: Bleeding on probing | From baseline (0 months) to follow-up (24 months)
  Change in proportion of bleeding sites on probing at baseline to follow-up (in percentage, %)
Response to treatment: Microbiological assay | From baseline (0 months) to follow-up (24 months)
  Change in proportion of specified microbes present in sample at baseline to follow-up
Response to treatment: GCF | From baseline (0 months) to follow-up (24 months)
  Change in proportion specified inflammatory markers present in sample at baseline to follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Nibali, PhD, Principal Investigator — Queen Mary University of London
Locations (2):
- United Kingdom (2):
  - Center for Oral Clinical Research, Queen Mary, University of London, London, Greater London
  - Dental and Maxillofacial Department, Great Ormond Street Hospital for Children, London

IPD SHARING:
Plan to Share IPD: No